CLINICAL TRIAL: NCT03672422
Title: Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC) CPDPC16-03 Pediatric Longitudinal Cohort Study of Chronic Pancreatitis
Brief Title: Pediatric Longitudinal Cohort Study of Chronic Pancreatitis
Acronym: INSPPIRE 2
Status: Completed | Type: Observational
Sponsor: Aliye Uc (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Aliye Uc, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201705709; 3U01DK108334 (NIH); NCT03081182 (obsolete NCT alias)
Record Dates: First submitted 2018-08-28; First posted 2018-09-14 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Pancreatitis, Chronic; Pancreatitis, Acute
Keywords: Pediatric; Pancreatitis; Chronic; Acute; Recurrent; ARP; CP; Pancreas; Children
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis; Bronchiolitis Obliterans Syndrome; Recurrence | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — 6 ml blood sample or 2 ml saliva sample collected 1 time. Urine 50 ml collected one time
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Recurrent Pancreatitis: At least 2 episodes of acute pancreatitis with complete resolution of pain and a >1 month pain-free interval between episodes.
  Interventions: Diagnostic Test: Blood sample; Behavioral: Patient questionnaires; Diagnostic Test: Saliva sample; Diagnostic Test: Urine sample
- Chronic Pancreatitis: Children with at least:
  1) One irreversible structural change* in the pancreas with or without abdominal pain +/- exocrine pancreatic insufficiency +/- diabetes.
  *irreversible structural changes:
  * Ductal calculi, dilated side branches, parenchymal calcifications found in any imaging (abdominal ultrasound (abd US), magnetic resonance imaging/magnetic resonance cholangiopancreatography (MRI/MRCP), computerized tomography (CT), endoscopic retrograde cholangiopancreatography (ERCP), endoscopic US (EUS).
  * Ductal obstruction or stricture/dilatation/irregularities that are persistent (for >2 months) on any imaging.
  * Parenchymal atrophy, irregular contour, accentuated lobular architecture, cavities alone are not diagnostic findings for CP.
  * Surgical or pancreatic biopsy specimen demonstrating histopathologic features compatible with CP (acinar atrophy, fibrosis, protein plugs, infiltration with lymphocytes, plasma cells, macrophages).
  Interventions: Diagnostic Test: Blood sample; Behavioral: Patient questionnaires; Diagnostic Test: Saliva sample; Diagnostic Test: Urine sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Six ml of blood will be collected from patients in an EDTA tube. 2 ml saliva samples in Oragene DNA collection kits
Behavioral: Patient questionnaires — Questionnaires will be completed at the baseline and annual follow-up visits to collect data that will define the demographics of the pediatric ARP and CP cohort, describe risk factors, presence of family history of acute and chronic pancreatitis, diabetes and pancreatic cancer and assess disease burden and sequelae.
Diagnostic Test: Saliva sample — 2 ml saliva samples in Oragene DNA collection kits collected if no blood sample being collected.
Diagnostic Test: Urine sample — 50 ml of urine in collection container.

SUMMARY:
The investigators will enroll a total of 628 patients under 18 years of age with ARP or CP. Included in the total are the 357patients in the INSPPIRE 1 database who are planned to be reenrolled under this protocol over the next 4 years. Patient questionnaires and physician surveys will be applied at the time of enrollment and annually thereafter as long as possible. At the first study visit after turning 18 years of age, the patient will sign the informed consent to continue in the study. Specifically, the investigators will define the demographics of the pediatric ARP and CP cohort, describe risk factors, presence of family history of acute and chronic pancreatitis, diabetes and pancreatic cancer and assess disease burden and sequelae.

DETAILED DESCRIPTION:
Disease Burden Pain. The pattern of the pain (constant versus episodic), its frequency, duration, visits to the emergency room or hospitalizations for pain, impact of pain on quality of life will be recorded in questionnaires. The intensity of the pain will be measured at enrollment, during an attack and annually using FACES Pain Scale-Revised, a self-report questionnaire validated for children >4 y/o. The names, dosing and frequency of medications taken for pain will also be queried.

Health-Related Quality of Life (HRQOL). An age-specific instrument validated for United States children will be used to measure HRQOL at enrollment and annually thereafter. Parents of children 5-18 years old will complete Child Health Questionnaire Parent Form 50 questions (CHQ PF-50). Children >10 years old will answer Child Health Questionnaire Child Form 87 questions (CHQ-87). Adults >18 years old will not complete a health-related questionnaire. These questionnaires capture physical functioning, social, emotional, physical and behavioral limitations, bodily pain, general behavior, mental health, self-esteem, general health perceptions, change in health and parental emotional impact.

Depression and anxiety. Depression and anxiety are strong predictors of chronic pain and pain-related disability in children, but it is not known whether this applies to children with ARP or CP. The investigators will assess for depression and anxiety in the INSPPIRE cohort at the time of enrollment and annually thereafter. The investigators will utilize the Child Behavioral Checklist (CBCL), one of the most widely-used standardized measures in child psychology for evaluating maladaptive behavioral and emotional problems in preschool subjects aged 1½ to 5 years and in school-age subjects between the ages of 6 and 18. For preschool-age children, the CBCL/1½-5 (completed by parents or surrogates) will be used. For school-age children 6-18 y/o, the investigators will utilize CBCL/6-18 y/o (completed by parents or surrogates). Children who are 11-18 y/o will answer a self-report questionnaire (Youth-Self Report Form or YSR/11-18). CBCL assesses internalizing (i.e., anxious, depressive, and over controlled) and externalizing (i.e., aggressive, hyperactive, noncompliant, and undercontrolled) behaviors. Adults >18 years old will not complete a behavioral checklist.

Patients/parents will spend approximately 2 hours answering questionnaires; their time will be compensated at $50 per visit. Patients will be enrolled during clinic visit as outpatient or as an inpatient. Alternatively, questionnaires can be applied over the phone or completed at home and returned via mail if the patient is unable to travel. Self-addressed stamped envelopes will be given to the patient/parent as needed for returning the questionnaires.

Disease Sequelae

The presence of exocrine pancreatic insufficiency and glucose intolerance/diabetes will be monitored at the time of enrollment and annually thereafter. Monitoring will include specifically:

1. Exocrine pancreatic insufficiency: defined as the presence of abnormal fecal elastase (< 100 ug/ g stool on 2 separate samples ≥ 1 month apart) or abnormal serum trypsin or serum trypsinogen.
2. Diabetes or prediabetes: Monitoring for diabetes in our cohort will include once yearly assessments with fasting glucose (diabetes range if ≥ 126 mg/dL), HbA1c (abnormal if >6; diabetic if >6.5%) and oral glucose tolerance test (OGTT). For OGTT, 1.75 grams/kg of standard glucose beverage (glucola, maximum 75 grams) will be consumed within 10 minutes at time 0. Glucose will be drawn prior to the beverage and at time 120 minutes. From this test, glycemic status will be defined as: (1) normal glucose tolerance (NGT, fasting glucose <100 mg/dL, 2 hour <140 mg/dL); (2) pre-diabetic based on impaired fasting glucose (IFG, fasting glucose 100-125 mg/dL) and/or impaired glucose tolerance (IGT, 2 hour glucose 140-199 mg/dL); or (3) diabetic (DM, fasting glucose >126 mg/dL or 2 hour glucose >200 mg/dL).
3. Nutritional status including micronutrient deficiency: To determine the nutritional sequelae of ARP or CP in children, the investigators will assess for malnutrition/obesity (weight, height, BMI, z scores; body fat mass and lean mass as measured by DXA scan), fat soluble vitamin deficiencies (serum vitamin levels for A, D, and E and bone density (DXA scan) in children with ARP or CP at the time of enrollment and annually thereafter.

The investigators will identify subjects within our cohort that presented with acute recurrent pancreatitis episodes, normal exocrine and endocrine pancreas function and normal pancreas imaging without any signs of chronicity (ARP cohort). The investigators will identify the development of CP on an annual basis as long as possible, as well as development of sequelae and disease burden as listed above.

Prospective Registry

The investigators will develop a database of children with ARP and CP. This will provide a cohort of well-phenotyped subjects for future studies targeting pathogenesis and novel therapies. The investigators will establish a process by which investigators outside of the consortium may have access to the data and biospecimens.

At enrollment, via the informed consent, subjects will choose whether or not to allow use of their biological samples for this study, future research, genetic analysis, genetic analysis for future research, and any type of future research. They will also choose whether or not we may keep their name and personal information in a registry to allow us to contact them for other future research.

BIOSPECIMEN COLLECTION

Sample collection for deoxyribonucleic acid (DNA): The subject will be able to give either blood or saliva. Six ml of blood will be collected from subjects in an ethylenediaminetetraacetic acid tube or 2 ml saliva samples in Oragene DNA collection kits then labeled with the barcoded specimen labels provided by the Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC) Coordinating Center. The specimen labels provided by CPDPC include a specimen identification (ID) number and barcode. Subject identifiers (for example names or initials) are not included on the labels. Before shipping the specimens to the central repository the specimen ID number from the label will be connected to the patient information in the CPDPC's secure IIMS Specimen Manager system. After the specimen ID number is linked to the subject in the CPDPC system the samples will be submitted to the central repository for the study via overnight courier. The central repository for DNA will be at the University of Iowa. The central repository at Iowa will not have access to the link that connects to the patient's personal identifiers in the Integrated Information Management System (IIMS). The central repository will log receipt of the specimens into the CPDPC IIMS Specimen Manager system using the specimen ID from the labeled vials. The central repository will process the specimens into aliquots for the extraction of genomic DNA following the CPDPC specimen processing described in the appendices. The aliquots will be labeled with CPDPC supplied labels and stored in a freezer at -80 degree Centigrade. The CPDPC aliquots labels contain barcodes and specimen ID numbers that do not link the aliquots to each other. The only link to the subject information resides in the secured database at the CPDPC coordinating and data management center. The central repository laboratory staff and the study researchers do not have access to this link. At the end of the study the specimens stored in the central repository at Iowa will be transferred to a central repository at National Institute of Diabetes and Digestive and Kidney Diseases.

Urine collection for bio-markers: To be completed only at sites identified by the lead site to collect urine samples. Not all sites will be collecting urine. See Appendix 14.27 for collection and processing instructions. The subject will be instructed to collect a minimum of 50 mL clean-catch urine sample. A dipstick urine analysis will be performed immediately after urine collection. Urine samples will then be kept on wet ice or refrigerated until processed. Samples will be processed within 4 hours of collection. Samples will be labeled with the barcoded specimen labels provided by the CPDPC Coordinating Center. The specimen labels provided by CPDPC include a specimen ID number and barcode. Subject identifiers (for example names or initials) are not included on the labels. Before shipping the specimens to the central repository the specimen ID number from the label will be connected to the subject information in the CPDPC's secure IIMS Specimen Manager system. After processing, samples will be frozen at -80ºC. The urine processing log sheet will be completed. Samples will be stored and batch shipped to the Central repository at University of Iowa annually. The central repository will log receipt of the specimens into the CPDPC IIMs Specimen Manager system using the specimen ID from the labeled vials. The central repository at University of Iowa will not have access to the link that connects the subject's personal identifiers in the IIMS system. The central repository will log receipt of the specimens into the CPDPC IIMS Specimen Manager system using the specimen ID from the labeled vials. The CPDPC aliquots labels contain barcodes and specimen ID numbers that do not link the aliquots to each other. The only link to the subject information resides in the secured database at the CPDPC coordinating and data management center. The central repository laboratory staff and the study researchers do not have access to this link. At the end of the study the specimens stored in the central repository at Iowa will be transferred to a central repository at NIDDK.

ELIGIBILITY:
Inclusion Criteria:

1. All patients/parents must sign an informed consent and/or assent indicating that they are aware of the investigational nature of this study.

2 Patients/parents must have signed an authorization for the release of their or their child's protected health information.

3 All children providing samples should fit the ARP or CP inclusion criteria defined below.

4 All children must be under 18 years of age at the time of enrollment.

Acute pancreatitis (AP): AP is defined as requiring 2 of the following:

1. Abdominal pain compatible with AP,
2. Serum amylase and/or lipase values ≥3 times upper limits of normal,
3. Imaging findings of AP, such as gland enlargement, acute inflammatory changes, and fluid collections.

ARP is defined as:

At least 2 episodes of acute pancreatitis with complete resolution of pain and a >1 month pain-free interval between episodes.

Chronic Pancreatitis:

Children with at least:

1. One irreversible structural change* in the pancreas with or without abdominal pain +/- exocrine pancreatic insufficiency +/- diabetes.

*irreversible structural changes:

* Ductal calculi, dilated side branches, parenchymal calcifications found in any imaging (abdominal ultrasound (abd US), magnetic resonance imaging/magnetic resonance cholangiopancreatography (MRI/MRCP), computerized tomography (CT), endoscopic retrograde cholangiopancreatography (ERCP), endoscopic US (EUS).
* Ductal obstruction or stricture/dilatation/irregularities that are persistent (for >2 months) on any imaging.
* Parenchymal atrophy, irregular contour, accentuated lobular architecture, cavities alone are not diagnostic findings for CP.
* Surgical or pancreatic biopsy specimen demonstrating histopathologic features compatible with CP (acinar atrophy, fibrosis, protein plugs, infiltration with lymphocytes, plasma cells, macrophages).

Exclusion Criteria:

* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate study interventions.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children <18 years of age with acute recurrent pancreatitis or chronic pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Length of time from progression from Acute Recurrent Pancreatitis to Chronic Pancreatitis | 3 years
  Date of diagnosis of first acute pancreatitis to date of diagnosis of chronic pancreatitis presented as minimum, maximum, median number of days and no progression to chronic pancreatitis.

SECONDARY OUTCOMES:
Number of subjects with abdominal pain | 1 year
  Presence of abdominal pain in the past year presented as number with "Yes", "No", "I don't know" and missing responses.
Number of subjects with constant abdominal pain | 1 year
  Presence of constant abdominal pain described as number of subjects with "Yes", "No", "I don't know" and missing responses.
Number of subjects with episodic abdominal pain | 1 year
  Number of subjects who are usually pain free with episodes of abdominal pain described as number with "Yes", "No", "I don't know" and missing responses..
Number of emergency room visits subject had in the past 12 months | 1 year
  Number of emergency room visits subjects experienced in the past 12 months presented as minimum, maximum, and median number of emergency room visits and number of missing responses.
Number of emergency room visits subject had in whole life | 18 years
  Number of emergency room visits the subject experienced in their whole life presented as minimum, maximum, and median number of visits and number of missing responses..
Number of hospitalizations subject had in past 12 months | 1 year
  Number of hospitalizations subject experienced in the past 12 months presented as minimum, maximum, and median number and number of missing responses..
Number of hospitalizations subject had in whole life | 18 years
  Number of hospitalizations subject had in their whole life presented as minimum, maximum, and median number and number of missing responses..
Number of school days subject missed in the last month | 30 days
  Number of school days subject missed in the last month presented as minimum, maximum, and median number and number of missing responses..
Number of subjects with Exocrine Pancreatic Insufficiency | 3 years
  Number of subjects with abnormal fecal elastase (< 100 micrograms/ gram of stool on 2 separate samples ≥ 1 month apart) presented as number of subjects with abnormal and normal lab values and number of subjects who did not have test done.
Number of subjects with abnormal fasting glucose | 3 years
  Number of subjects with fasting glucose ≥126 milligrams per deciliter presented as number of subjects with abnormal and normal lab value and number of subjects who did not have test done.
Number of subjects with abnormal hemoglobin A1c (HbA1c) | 3 years
  Number of subjects with HbA1c (abnormal if >6; diabetic if >6.5%) results that were normal, abnormal, and diabetic and number who did not have test done.
Number of subjects with abnormal oral glucose tolerance test (OGTT) | 3 years
  Number of subjects with abnormal OGTT test results. OGTT performed with 1.75 grams/kilogram of standard glucose beverage (glucola, maximum 75 grams) consumed within 10 minutes at time 0. Glucose drawn prior to the beverage and at time 120 minutes. Glycemic status will be defined as: (1) normal glucose tolerance (NGT, fasting glucose <100 mg/dL, 2 hour <140 mg/dL); (2) pre-diabetic based on impaired fasting glucose (IFG, fasting glucose 100-125 mg/dL) and/or impaired glucose tolerance (IGT, 2 hour glucose 140-199 mg/dL); or (3) diabetic (DM, fasting glucose >126 mg/dL or 2 hour glucose >200 mg/dL). Findings presented as number of subjects with normal, pre-diabetic, impaired, and diabetic results and number that did not have test done.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Ph.D, Study Director — MD Anderson
Locations (22):
- United States (18):
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Riley Hospital for Children Indiana University, Indianapolis, Indiana
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philipsburg, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Health University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Sydney Children's Hospital Randwick, Randwick, New South Wales, Australia
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Hadassah University Hospital Mt. Scopus, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu-El-Haija M, Kumar S, Quiros JA, Balakrishnan K, Barth B, Bitton S, Eisses JF, Foglio EJ, Fox V, Francis D, Freeman AJ, Gonska T, Grover AS, Husain SZ, Kumar R, Lapsia S, Lin T, Liu QY, Maqbool A, Sellers ZM, Szabo F, Uc A, Werlin SL, Morinville VD. Management of Acute Pancreatitis in the Pediatric Population: A Clinical Report From the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition Pancreas Committee. J Pediatr Gastroenterol Nutr. 2018 Jan;66(1):159-176. doi: 10.1097/MPG.0000000000001715. PMID 29280782
- [Background] Abu-El-Haija M, Uc A, Werlin SL, Freeman AJ, Georgieva M, Jojkic-Pavkov D, Kalnins D, Kochavi B, Koot BGP, Van Biervliet S, Walkowiak J, Wilschanski M, Morinville VD. Nutritional Considerations in Pediatric Pancreatitis: A Position Paper from the NASPGHAN Pancreas Committee and ESPGHAN Cystic Fibrosis/Pancreas Working Group. J Pediatr Gastroenterol Nutr. 2018 Jul;67(1):131-143. doi: 10.1097/MPG.0000000000002023. PMID 29927872
- [Background] Morinville VD, Husain SZ, Bai H, Barth B, Alhosh R, Durie PR, Freedman SD, Himes R, Lowe ME, Pohl J, Werlin S, Wilschanski M, Uc A; INSPPIRE Group. Definitions of pediatric pancreatitis and survey of present clinical practices. J Pediatr Gastroenterol Nutr. 2012 Sep;55(3):261-5. doi: 10.1097/MPG.0b013e31824f1516. PMID 22357117
- [Background] Morinville VD, Lowe ME, Ahuja M, Barth B, Bellin MD, Davis H, Durie PR, Finley B, Fishman DS, Freedman SD, Gariepy CE, Giefer MJ, Gonska T, Heyman MB, Himes R, Husain S, Kumar S, Ooi CY, Pohl JF, Schwarzenberg SJ, Troendle D, Werlin SL, Wilschanski M, Yen E, Uc A. Design and implementation of INSPPIRE. J Pediatr Gastroenterol Nutr. 2014 Sep;59(3):360-4. doi: 10.1097/MPG.0000000000000417. PMID 24824361
- [Background] Perito ER, Rhee S. Relief for Young Children With Severe Chronic Pancreatitis. J Pediatr Gastroenterol Nutr. 2017 Mar;64(3):338-339. doi: 10.1097/MPG.0000000000001509. No abstract available. PMID 28231070
- [Background] Uc A, Andersen DK, Bellin MD, Bruce JI, Drewes AM, Engelhardt JF, Forsmark CE, Lerch MM, Lowe ME, Neuschwander-Tetri BA, O'Keefe SJ, Palermo TM, Pasricha P, Saluja AK, Singh VK, Szigethy EM, Whitcomb DC, Yadav D, Conwell DL. Chronic Pancreatitis in the 21st Century - Research Challenges and Opportunities: Summary of a National Institute of Diabetes and Digestive and Kidney Diseases Workshop. Pancreas. 2016 Nov;45(10):1365-1375. doi: 10.1097/MPA.0000000000000713. PMID 27748719
- [Background] Uc A, Fishman DS. Pancreatic Disorders. Pediatr Clin North Am. 2017 Jun;64(3):685-706. doi: 10.1016/j.pcl.2017.01.010. PMID 28502446
- [Result] Gariepy CE, Heyman MB, Lowe ME, Pohl JF, Werlin SL, Wilschanski M, Barth B, Fishman DS, Freedman SD, Giefer MJ, Gonska T, Himes R, Husain SZ, Morinville VD, Ooi CY, Schwarzenberg SJ, Troendle DM, Yen E, Uc A. Causal Evaluation of Acute Recurrent and Chronic Pancreatitis in Children: Consensus From the INSPPIRE Group. J Pediatr Gastroenterol Nutr. 2017 Jan;64(1):95-103. doi: 10.1097/MPG.0000000000001446. PMID 27782962
- [Result] Giefer MJ, Lowe ME, Werlin SL, Zimmerman B, Wilschanski M, Troendle D, Schwarzenberg SJ, Pohl JF, Palermo J, Ooi CY, Morinville VD, Lin TK, Husain SZ, Himes R, Heyman MB, Gonska T, Gariepy CE, Freedman SD, Fishman DS, Bellin MD, Barth B, Abu-El-Haija M, Uc A. Early-Onset Acute Recurrent and Chronic Pancreatitis Is Associated with PRSS1 or CTRC Gene Mutations. J Pediatr. 2017 Jul;186:95-100. doi: 10.1016/j.jpeds.2017.03.063. Epub 2017 May 10. PMID 28502372
- [Result] Husain SZ, Morinville V, Pohl J, Abu-El-Haija M, Bellin MD, Freedman S, Hegyi P, Heyman MB, Himes R, Ooi CY, Schwarzenberg SJ, Usatin D, Uc A. Toxic-metabolic Risk Factors in Pediatric Pancreatitis: Recommendations for Diagnosis, Management, and Future Research. J Pediatr Gastroenterol Nutr. 2016 Apr;62(4):609-17. doi: 10.1097/MPG.0000000000001035. PMID 26594832
- [Result] Kumar S, Ooi CY, Werlin S, Abu-El-Haija M, Barth B, Bellin MD, Durie PR, Fishman DS, Freedman SD, Gariepy C, Giefer MJ, Gonska T, Heyman MB, Himes R, Husain SZ, Lin TK, Lowe ME, Morinville V, Palermo JJ, Pohl JF, Schwarzenberg SJ, Troendle D, Wilschanski M, Zimmerman MB, Uc A. Risk Factors Associated With Pediatric Acute Recurrent and Chronic Pancreatitis: Lessons From INSPPIRE. JAMA Pediatr. 2016 Jun 1;170(6):562-9. doi: 10.1001/jamapediatrics.2015.4955. PMID 27064572
- [Result] Lin TK, Abu-El-Haija M, Nathan JD, Palermo JP, Barth B, Bellin M, Fishman DS, Freedman SD, Gariepy CE, Giefer MJ, Gonska T, Heyman MB, Himes R, Husain SZ, Liu Q, Maqbool A, Mascarenhas M, McFerron B, Morinville VD, Ooi CY, Perito E, Pohl JF, Rhee S, Schwarzenberg SJ, Shah U, Troendle D, Werlin SL, Wilschanski M, Zimmerman MB, Lowe ME, Uc A. Pancreas Divisum in Pediatric Acute Recurrent and Chronic Pancreatitis: Report From INSPPIRE. J Clin Gastroenterol. 2019 Jul;53(6):e232-e238. doi: 10.1097/MCG.0000000000001063. PMID 29864067
- [Result] Pohl J, Morinville V, Husain SZ, Uc A. Toxic-Metabolic Risk Factors Are Uncommon in Pediatric Chronic Pancreatitis. J Pediatr Gastroenterol Nutr. 2016 Jun;62(6):e66-7. doi: 10.1097/MPG.0000000000001156. No abstract available. PMID 27213250
- [Result] Scheers I, Palermo JJ, Freedman S, Wilschanski M, Shah U, Abu-El-Haija M, Barth B, Fishman DS, Gariepy C, Giefer MJ, Heyman MB, Himes RW, Husain SZ, Lin TK, Liu Q, Lowe M, Mascarenhas M, Morinville V, Ooi CY, Perito ER, Piccoli DA, Pohl JF, Schwarzenberg SJ, Troendle D, Werlin S, Zimmerman B, Uc A, Gonska T. Recommendations for Diagnosis and Management of Autoimmune Pancreatitis in Childhood: Consensus From INSPPIRE. J Pediatr Gastroenterol Nutr. 2018 Aug;67(2):232-236. doi: 10.1097/MPG.0000000000002028. PMID 29746340
- [Result] Troendle DM, Fishman DS, Barth BA, Giefer MJ, Lin TK, Liu QY, Abu-El-Haija M, Bellin MD, Durie PR, Freedman SD, Gariepy C, Gonska T, Heyman MB, Himes R, Husain SZ, Kumar S, Lowe ME, Morinville VD, Ooi CY, Palermo J, Pohl JF, Schwarzenberg SJ, Werlin S, Wilschanski M, Zimmerman MB, Uc A. Therapeutic Endoscopic Retrograde Cholangiopancreatography in Pediatric Patients With Acute Recurrent and Chronic Pancreatitis: Data From the INSPPIRE (INternational Study group of Pediatric Pancreatitis: In search for a cuRE) Study. Pancreas. 2017 Jul;46(6):764-769. doi: 10.1097/MPA.0000000000000848. PMID 28609364
- [Result] Scheers I, Palermo JJ, Freedman S, Wilschanski M, Shah U, Abu-El-Haija M, Barth B, Fishman DS, Gariepy C, Giefer MJ, Heyman MB, Himes RW, Husain SZ, Lin TK, Liu Q, Lowe M, Mascarenhas M, Morinville V, Ooi CY, Perito ER, Piccoli DA, Pohl JF, Schwarzenberg SJ, Troendle D, Werlin S, Zimmerman B, Uc A, Gonska T. Autoimmune Pancreatitis in Children: Characteristic Features, Diagnosis, and Management. Am J Gastroenterol. 2017 Oct;112(10):1604-1611. doi: 10.1038/ajg.2017.85. Epub 2017 Apr 4. PMID 28374818
- [Result] Schwarzenberg SJ, Bellin M, Husain SZ, Ahuja M, Barth B, Davis H, Durie PR, Fishman DS, Freedman SD, Gariepy CE, Giefer MJ, Gonska T, Heyman MB, Himes R, Kumar S, Morinville VD, Lowe ME, Nuehring NE, Ooi CY, Pohl JF, Troendle D, Werlin SL, Wilschanski M, Yen E, Uc A. Pediatric chronic pancreatitis is associated with genetic risk factors and substantial disease burden. J Pediatr. 2015 Apr;166(4):890-896.e1. doi: 10.1016/j.jpeds.2014.11.019. Epub 2014 Dec 30. PMID 25556020
- [Result] Ting J, Wilson L, Schwarzenberg SJ, Himes R, Barth B, Bellin MD, Durie PR, Fishman DS, Freedman SD, Gariepy CE, Giefer MJ, Gonska T, Husain SZ, Kumar S, Morinville VD, Lowe ME, Ooi CY, Pohl JF, Troendle D, Usatin D, Werlin SL, Wilschanski M, Heyman MB, Uc A. Direct Costs of Acute Recurrent and Chronic Pancreatitis in Children in the INSPPIRE Registry. J Pediatr Gastroenterol Nutr. 2016 Mar;62(3):443-9. doi: 10.1097/MPG.0000000000001057. PMID 26704866
- See also: INSPPIRE Pediatric Pancreatitis Research Project — https://medicine.uiowa.edu/pediatrics/research/insppire-pediatric-pancreatitis-research-project